CLINICAL TRIAL: NCT04897672
Title: Use of 2D-Speckle Tracking Echocardiography in a Pediatric Population With Chronic Renal Disease: a Multicentre Cross-sectional Controlled Study (SPECKLE-KIDNEY-PED)
Brief Title: 2D-speckle Tracking in Pediatric Renal Chronic Disease
Acronym: SPECKLEKIDNEY
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); University Hospital, Limoges (Other); Marseille University Hospital- La Timone (Unknown); Hopital Universitaire Robert-Debre (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0344
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic Renal Disease; Chronic Renal Insufficiency; Congenital Heart Disease
Keywords: Speckle-tracking; Exercice capacity; Cardiovascular prognosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Defects, Congenital | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: case: Children aged 6 to 17 years old reffered to the pediatric cardiology consultation with a chronic renal disease and renal insufficiency
  Interventions: Other: Observational study
- control: control : Children aged 6 to 17 years old reffered to the pediatric cardiology consultation who were classified in the control group after a completely normal check-up, including physical examination, electrocardiogram, and echocardiography
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
The SPECKLE- KIDNEY-PED is a multicentre observational controlled trial aiming to evaluate the 2D-Speckle tracking in a population of 85 patients aged from 6 to 17 years old with a chronic renal disease and to compare the results to those of 85 age and gender-matched healthy subjects. The secondary objective is to assess the conventional echocardiographic parameters and the level of exercice capacity.

DETAILED DESCRIPTION:
Kidney disease and chronic kidney failure are one of the most common causes of chronic childhood disease. They are often complicated by cardiovascular disease, which can, in the long run, affect patients' prognosis. Thus, mortality in children undergoing hemodialysis for end-stage kidney failure is related in more than 30% of cases to a cardiovascular complication. An annual cardiac assessment is recommended as part of the follow-up of these patients to assess the cardiac impact of kidney disease (high blood pressure, hyper-uremia, etc.). The use of conventional cardiological assessment parameters does not predict the cardiovascular prognosis of patients because the alteration of these parameters is greatly delayed in the course of the disease. 2D strain or "speckle tracking echocardiography" is a non-invasive ultrasound technique that allows for a more sensitive assessment of myocardial tissue damage and its early impairment has been shown as a factor of poor prognosis in other pediatric chronic pathology (neuromuscular disease, cardiotoxic exposure, etc.) as well as in adult chronic kidney failure.

The SPECKLE- KIDNEY-PED trial is a multicentre observationnal controlled study. The main objective of this work is to asses the 2D strain ventricular function in children with kidney failure, to compare it with that of healthy children of 6 to 17 years old, and to correlate it with the cardio-renal severity of the disease in terms of level of kidney failure and aerobic physical fitness.

The secondary objective is to assess, in this population, the level of exercice capacity and to compare it to the general population of children of the same age.

A total of 180 children are recquired to observe a significant difference of 2,5% of the global strain value with a power of 90% and an alpha risk of 5%.

The SPECKLE- KIDNEY-PED trial intends to improve the level of evidence for future guidelines on cardiologic survey and promotion of physical activity in this population

ELIGIBILITY:
Inclusion criteria:

* Patient aged 6 to 17 years old
* Patient with chronic renal disease (>3 months)
* Patient with renal insufficiency (glomerular filtration rate < 80ml/min/1,73m2)

Exclusion criteria:

* Patient with associated congenital heart disease
* Patient with uncontrolled arrythmia

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases group : Children aged 6 to 17years old with chronic renal insufficiency
  Control group: Children aged 6 to 17 years old with normal check up
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Global and segmentary longitudinal 2D- speckle tracking value of the left ventricule by transthoracic echocardiography | Baseline (1day)
  Transthoracic echocardiography parameters

SECONDARY OUTCOMES:
Conventional echocardiography parameters | Baseline (1day)
  ransthoracic echocardiography parameters
Exercice capacity | Baseline (1day)
  Cardiopulmonary exercice test with VO2max assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER; Oscar WERNER, MD, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC